CLINICAL TRIAL: NCT00146055
Title: Low-Intensity Preparative Regimen and Allogeneic Peripheral Blood Stem Cell Transplantation From Unrelated Donor in Patients With Hematologic Malignancy
Brief Title: Low-Intensity Preparation and Allogeneic Transplant in Patients With Cancers of the Blood
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 9970
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Myeloma, Plasma-Cell; Lymphoma, Malignant; Myeloproliferative Disorders; Myelodysplastic Syndromes; Waldenstrom's Macroglobulinemia
MeSH Terms: conditions — Multiple Myeloma; Lymphoma; Myeloproliferative Disorders; Myelodysplastic Syndromes; Waldenstrom Macroglobulinemia | interventions — Transplantation, Homologous

INTERVENTIONS:
Procedure: Reduced intensity conditioning with allogeneic transplant

SUMMARY:
The purpose of this study is to determine whether a less-intensive preparative therapy followed by an allogeneic peripheral stem cell transplantation will provide an effective treatment for your disease and whether it will be associated with fewer side effects.

DETAILED DESCRIPTION:
Combinations of high-dose chemotherapy and radiation therapy (preparative regimen) followed with allogeneic bone marrow or stem cell transplantation from an unrelated donor is a current treatment approach. Chemotherapeutic drugs and radiation are given in higher doses to increase their effectiveness. High-dose chemotherapy and radiation therapy generally affect cells that are dividing. They are used to treat cancer because cancer cells divide more often than most other cells. High-dose treatment severely damages the patient's bone marrow so that the patient no longer is able to produce needed blood cells. Peripheral stem cell transplantation allows stem cells that were damaged by treatment to be replaced with healthy stem cells that can produce the blood cells the patient needs. Patients experience a number of complications after transplantation. Some are temporary and relatively minor; yet others can be life threatening. Many doctors consider high-dose chemotherapy, by itself or with radiation, and bone marrow or stem cell transplantation as the best available treatment option for diseases under specific circumstances. However, this study will explore whether a less-intensive preparative therapy before the peripheral stem cell transplantation will prove to be safer, have less side effects, and be an effective treatment for certain diseases.

ELIGIBILITY:
Inclusion Criteria:

Patients must be a candidate for unrelated donor stem cell transplantation and the donor and recipient must be 5/6 or 6/6 matched. In addition, patients must have one of the following histologically confirmed diagnosis :

1. Patients with previously treated AML (M0 - M7 by FAB classification)

   * who are in not in complete remission (CR).
   * who are in second or later CR.
   * who have 5-30% persistent blasts in bone marrow following induction or salvage chemotherapy.
   * who have high-risk feature in first complete remission e.g. presence of Philadelphia chromosome or non-core-binding factor type of chromosomal abnormalities.
2. Patients with myelodysplastic syndromes and IPS int-1, int-2 or high-risk scores who are transfusion-dependent.
3. Patients with chronic myeloid leukemia who are in accelerated, blastic, or or chronic phase
4. Patients with acute lymphoblastic leukemia

   * who are in first complete remission and have high risk disease [Ph' or t (4; 11) , WBC> 30,000, > 4 weeks to achieve CR].
   * who are in second or greater CR.
   * who did not achieve a CR following induction or salvage therapy.
5. Patients with Hodgkin's or non-Hodgkin's lymphoma who are not curable with conventional chemotherapy and do not have any tumor larger than 5 centimeters in diameter.
6. Patients with myeloma or plasma cell neoplasms who are :

   * stage III at presentation.
   * stage I-II at presentation but were not responding or progressed after first line therapy.
7. Patient with chronic lymphocytic leukemia or Waldenström's macroglobulinemia who progressed after first-line therapy.
8. Patients with MDS or myeloproliferative disorders who had history of life-threatening complications related to thrombosis, hemorrhagic diathesis or intractable hypercatabolic state (fever cachexia).

Exclusion Criteria:

1. Cardiac disease of symptomatic nature; < 25% ejection fraction.
2. Severe renal disease; creatinine > 2.O mg/dl or creatinine clearance < 40 ml/min. (Corrected for age)
3. Severe pulmonary disease < 60% normal (FEV1 & FVC).
4. Severe hepatic disease; bilirubin >2.0, and/or transaminase > 3 x normal corrected for age.
5. Karnofsky performance status of < 60%.
6. Patients with evidence of HIV infection by western blot.
7. Any conditions, in the opinion of the transplant team such as substance abuse, or severe personality disorder that would keep the patients from complying with the needs of the protocol and would markedly increase the morbidity and mortality from the procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2000-03; Primary Completion 2004-11 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
- To evaluate the toxicity of low-intensity regimen for allogeneic stem cell transplantation from an unrelated donor.
- To evaluate the engraftment, and chimerism.
- To estimate the rate of acute GVHD, relapse and survival.

CONTACTS AND LOCATIONS:
Overall Officials: John E. Levine, MS MD, Principal Investigator — The Univeristy of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States